CLINICAL TRIAL: NCT05161975
Title: Effects of Vitamin K2 Supplements on Recovery of Lower Limb Muscle Function After Ankle Injury in Adults
Brief Title: Vitamin K2 Supplements for Muscle Recovery
Acronym: Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lithuanian Sports University (Other)
Collaborators: Kappa Bioscience AS (Unknown); LSMU Kauno ligonine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LithuanianSportsU-7
Record Dates: First submitted 2021-11-11; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Muscle Atrophy; Cachexia
Keywords: Cachexia; Insulin Resistance; Muscle Weakness; Exercise training
MeSH Terms: conditions — Muscular Atrophy; Cachexia; Insulin Resistance; Muscle Weakness | interventions — Vitamin K 2

STUDY DESIGN:
Intervention Model Description: We will carry out a double-blinded, randomized, placebo controlled clinical trial. We will recruit 18-60 years old men and women who have sustained ankle injury and arrived to LSMU Kauno ligonine for treatment. The volunteers will be randomly assigned to the vitamin K2 (MK-7, 330 micrograms) or placebo group. We expect to see 3-mm difference in muscle thickness between the groups. The gastrocnemius muscle thickness is reported to be 17.49 ± 3.81 mm (Kirmaci et al. 2021). Thus, 25 volunteers in each group are needed (statistical power = 80%, p < 0.05) for the study. We will recruit 30 volunteers into each group as some volunteers might drop out of the study. We will recruit equal number of 18-39 year old and 40-59 year olds into both groups (n =15 each) to minimize effects of age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Food supplement tablets do not contain vitamin K2
  Interventions: Dietary Supplement: Vitamin K2
- Vitamin K2 (Experimental): Food supplement tablets contain vitamin K2
  Interventions: Dietary Supplement: Vitamin K2

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — Volunteers will be randomly assigned to vitamin K2 or placebo group and consume one tablet of the food supplement per day.

SUMMARY:
Ankle injury is one of the most common injuries which can have long term consequences. Ankle immobilization is often applied for up to six weeks to ensure healing of the soft tissue and fractured bones after such an injury. This causes significant wasting of the lower leg muscles driven by inflammation and oxidative stress. The rate of muscle atrophy and recovery after injury varies significantly by sex and age. These differences might be linked to changes in gene and protein expression associated with regulation of protein synthesis and proteolysis. Interventions that reduce the deleterious effects of ankle injury as well as understanding of the underlying mechanisms could be particularly useful in promotion of healthy ageing. Vitamin K includes a group of structurally related compounds. Phylloquinone (vitamin K1) and menaquinones (vitamin K2s) of which MK-4 and MK-7 are the most important. Vitamin K2 has anti-inflammatory and antioxidant effects and thus may be effective in reducing muscle atrophy during limb immobilization and improving recovery of muscle function after injury. This aim of the current study is to investigate if vitamin K2 supplements can ameliorate muscle atrophy and improve recovery of muscle function after ankle injury. The investigators will study younger (18-39 year old) and older (40-60 year old) men and women to assess effects of sex and age.

DETAILED DESCRIPTION:
Muscle weakness is associated with impaired quality of life, increased risk of falling, disability and premature mortality. Whilst ageing results in a progressive decline, even short periods of low physical activity can result in significant deterioration of muscle function and metabolic health. One such period of very low activity can occur following illness or injury. This can lead to decrease in lower limb muscle mass and strength. Muscle exercise training promotes recovery of skeletal muscles after injury though improvements vary between individuals and appear to decrease with age. Strategies to retard loss of muscle mass and function during inactivity are, thus, of critical importance in understanding of the mechanisms underlying such effects.

Vitamin K includes a group of structurally related compounds named phylloquinone (vitamin K1) and menaquinones (vitamin K2s) of which MK-4 and MK-7 are the most important. Vitamin K is an essential cofactor for gamma carboxylation, required for the effective function of a range of proteins and has been linked to chronic disease and inflammation. Muscle cell studies suggest that vitamin K2 increases expression of myogenic transcription factors such as MyoD and promotes muscle cell proliferation. There are 20 described vitamin K dependent proteins (VKDPs). It is also known that vitamin K2 inhibits the activation of NFkB independently of gamma-carboxylation. This prevents nuclear entry of NFkB and therefore, consequently, vitamin K2 inhibits NFkB to interact with its nuclear receptors. In addition, Vitamin K2 can function as an electron carrier in mitochondria, and therefore play an inhibitory role on oxidative stress and release of ROS. There is, therefore, a strong rationale for investigating the effects of vitamin K2 during ankle immobilisation. The aim of the study is to investigate the effects of vitamin K2 on skeletal muscles after ankle injury and in the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age;
* Lives in Lithuania;
* Able and willing to give informed written consent to participate in the study;
* Recent (24 h before volunteering for the study) ankle injury requiring 6-week ankle immobilization;
* Exercise training program during 6-week recovery is recommended.

Exclusion Criteria:

* Body mass index (BMI) is greater than 30 kg / m2;
* Diabetes complicates cardiovascular diseases,
* Liver disease;
* Blood pressure is greater than 150/90mmHg during the first measurement;
* Incidences of consciousness loss;
* Cancer;
* Dementia;
* Other injuries that affect lower limb muscles;
* Use of anticoagulant drugs;
* Smoking;
* Drug abuse;
* Using drugs that affect muscle function (steroids).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | 12 weeks.
  Transverse images of medial and lateral gastrocnemius, soleus and tibialis anterior muscles will be obtained using B-mode ultrasonography with a 10-15 MHz transducer.
Muscle strength | 12 weeks.
  Plantar flexor and extensor strength will be measured using isokinetic dynamometer (Biodex System 3 Biodex Medical Systems, Inc., Shirley, NY, USA).
Vitamin K2 status | 12 weeks.
  Blood samples will be taken and plasma levels of vitamin K2 will be assessed.

SECONDARY OUTCOMES:
Cytokine profile | 12 weeks.
  Blood samples will be taken and ELISA assays for insulin, myostatin, TGF-β2, IGF-1, IL-1b, IL-6 and TNF-alpha will be performed
Gene expression profile | 12 weeks.
  Biopsies of soleus and gastrocnemius muscles will be taken. The mRNA levels of p62, Atrogin 1, MuRF 1, LC3b and Gapdh were assessed using SYBR Green (#4367659, Thermo Fisher Scientific) assay for quantitative PCR.
Protein expression profile | 12 weeks.
  Biopsies of soleus and gastrocnemius muscles will be taken. Western blotting will be carried to examine signalling pathways that control protein synthase (Akt-mTOR-p70s6k).
Metabolic enzyme activity | 12 weeks.
  Biopsies of soleus and gastrocnemius muscles will be taken. Enzyme assays for citrate synthase (CS), succinate dehydrogenase (SDH), β-hydroxyacyl-coenzyme dehydrogenase (HAD) and other metabolic enzyme will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Aivaras Ratkevicius, Dr., Principal Investigator — Lithuanian Sports University
Locations (2):
- Lithuania (2):
  - Lithuanian Sports University, Kaunas
  - LSMU Kauno ligonine, Kaunas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe RR. The underappreciated role of muscle in health and disease. Am J Clin Nutr. 2006 Sep;84(3):475-82. doi: 10.1093/ajcn/84.3.475. PMID 16960159
- [Background] Celis-Morales CA, Welsh P, Lyall DM, Steell L, Petermann F, Anderson J, Iliodromiti S, Sillars A, Graham N, Mackay DF, Pell JP, Gill JMR, Sattar N, Gray SR. Associations of grip strength with cardiovascular, respiratory, and cancer outcomes and all cause mortality: prospective cohort study of half a million UK Biobank participants. BMJ. 2018 May 8;361:k1651. doi: 10.1136/bmj.k1651. PMID 29739772
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Krogh-Madsen R, Thyfault JP, Broholm C, Mortensen OH, Olsen RH, Mounier R, Plomgaard P, van Hall G, Booth FW, Pedersen BK. A 2-wk reduction of ambulatory activity attenuates peripheral insulin sensitivity. J Appl Physiol (1985). 2010 May;108(5):1034-40. doi: 10.1152/japplphysiol.00977.2009. Epub 2009 Dec 31. PMID 20044474
- [Background] Juto H, Nilsson H, Morberg P. Epidemiology of Adult Ankle Fractures: 1756 cases identified in Norrbotten County during 2009-2013 and classified according to AO/OTA. BMC Musculoskelet Disord. 2018 Dec 13;19(1):441. doi: 10.1186/s12891-018-2326-x. PMID 30545314
- [Background] Psatha M, Wu Z, Gammie FM, Ratkevicius A, Wackerhage H, Lee JH, Redpath TW, Gilbert FJ, Ashcroft GP, Meakin JR, Aspden RM. A longitudinal MRI study of muscle atrophy during lower leg immobilization following ankle fracture. J Magn Reson Imaging. 2012 Mar;35(3):686-95. doi: 10.1002/jmri.22864. Epub 2011 Nov 1. PMID 22045592
- [Background] Stevens JE, Pathare NC, Tillman SM, Scarborough MT, Gibbs CP, Shah P, Jayaraman A, Walter GA, Vandenborne K. Relative contributions of muscle activation and muscle size to plantarflexor torque during rehabilitation after immobilization. J Orthop Res. 2006 Aug;24(8):1729-36. doi: 10.1002/jor.20153. PMID 16779833
- [Background] Psatha M, Wu Z, Gammie F, Ratkevicius A, Wackerhage H, Redpath TW, Gilbert FJ, Meakin JR, Aspden RM. Age-related changes in the effects of strength training on lower leg muscles in healthy individuals measured using MRI. BMJ Open Sport Exerc Med. 2017 Jul 20;3(1):e000249. doi: 10.1136/bmjsem-2017-000249. eCollection 2017. PMID 28761720
- [Background] Rosa-Caldwell ME, Lim S, Haynie WS, Jansen LT, Westervelt LC, Amos MG, Washington TA, Greene NP. Altering aspects of mitochondrial quality to improve musculoskeletal outcomes in disuse atrophy. J Appl Physiol (1985). 2020 Dec 1;129(6):1290-1303. doi: 10.1152/japplphysiol.00407.2020. Epub 2020 Sep 17. PMID 32940556
- [Background] Sitnick M, Bodine SC, Rutledge JC. Chronic high fat feeding attenuates load-induced hypertrophy in mice. J Physiol. 2009 Dec 1;587(Pt 23):5753-65. doi: 10.1113/jphysiol.2009.180174. Epub 2009 Oct 12. PMID 19822547
- [Background] Hotamisligil GS. Foundations of Immunometabolism and Implications for Metabolic Health and Disease. Immunity. 2017 Sep 19;47(3):406-420. doi: 10.1016/j.immuni.2017.08.009. PMID 28930657
- [Background] Laufs U, Wassmann S, Czech T, Munzel T, Eisenhauer M, Bohm M, Nickenig G. Physical inactivity increases oxidative stress, endothelial dysfunction, and atherosclerosis. Arterioscler Thromb Vasc Biol. 2005 Apr;25(4):809-14. doi: 10.1161/01.ATV.0000158311.24443.af. Epub 2005 Feb 3. PMID 15692095
- [Background] Meng SJ, Yu LJ. Oxidative stress, molecular inflammation and sarcopenia. Int J Mol Sci. 2010 Apr 12;11(4):1509-26. doi: 10.3390/ijms11041509. PMID 20480032
- [Background] Atherton PJ, Greenhaff PL, Phillips SM, Bodine SC, Adams CM, Lang CH. Control of skeletal muscle atrophy in response to disuse: clinical/preclinical contentions and fallacies of evidence. Am J Physiol Endocrinol Metab. 2016 Sep 1;311(3):E594-604. doi: 10.1152/ajpendo.00257.2016. Epub 2016 Jul 5. PMID 27382036
- [Background] Shearer MJ, Okano T. Key Pathways and Regulators of Vitamin K Function and Intermediary Metabolism. Annu Rev Nutr. 2018 Aug 21;38:127-151. doi: 10.1146/annurev-nutr-082117-051741. Epub 2018 Jun 1. PMID 29856932
- [Background] Harshman SG, Shea MK. The Role of Vitamin K in Chronic Aging Diseases: Inflammation, Cardiovascular Disease, and Osteoarthritis. Curr Nutr Rep. 2016 Jun;5(2):90-98. doi: 10.1007/s13668-016-0162-x. Epub 2016 Mar 31. PMID 27648390
- [Background] Haugsgjerd TR, Egeland GM, Nygard OK, Vinknes KJ, Sulo G, Lysne V, Igland J, Tell GS. Association of dietary vitamin K and risk of coronary heart disease in middle-age adults: the Hordaland Health Study Cohort. BMJ Open. 2020 May 21;10(5):e035953. doi: 10.1136/bmjopen-2019-035953. PMID 32444431
- [Background] Azuma K, Inoue S. Multiple Modes of Vitamin K Actions in Aging-Related Musculoskeletal Disorders. Int J Mol Sci. 2019 Jun 11;20(11):2844. doi: 10.3390/ijms20112844. PMID 31212662
- [Background] Ronning SB, Pedersen ME, Berg RS, Kirkhus B, Rodbotten R. Vitamin K2 improves proliferation and migration of bovine skeletal muscle cells in vitro. PLoS One. 2018 Apr 4;13(4):e0195432. doi: 10.1371/journal.pone.0195432. eCollection 2018. PMID 29617432
- [Background] Simes DC, Viegas CSB, Araujo N, Marreiros C. Vitamin K as a Powerful Micronutrient in Aging and Age-Related Diseases: Pros and Cons from Clinical Studies. Int J Mol Sci. 2019 Aug 25;20(17):4150. doi: 10.3390/ijms20174150. PMID 31450694
- [Background] McGlory C, Gorissen SHM, Kamal M, Bahniwal R, Hector AJ, Baker SK, Chabowski A, Phillips SM. Omega-3 fatty acid supplementation attenuates skeletal muscle disuse atrophy during two weeks of unilateral leg immobilization in healthy young women. FASEB J. 2019 Mar;33(3):4586-4597. doi: 10.1096/fj.201801857RRR. Epub 2019 Jan 10. PMID 30629458